CLINICAL TRIAL: NCT03504332
Title: Clinical and Radiographic Evaluation of Calcium Hydroxide and Bi-antibiotic Paste as Anti-microbial Dressing in Revascularization of Non Vital Immature Permanent Anterior Teeth: A Randomized Clinical Trial
Brief Title: Revascularization of Immature Anterior Necrotic Teeth
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohamed Fouad Wahby, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: regenerative endodontics
Record Dates: First submitted 2018-04-05; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Pulp Necroses
Keywords: immature teeth, revascularization
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxide in revascularization (Experimental): Revascularization of necrotic anterior teeth: canals disinfection step. Pure Calcium Hydroxide powder mixed with saline will be placed as intra-canal medication in the 1st visit of dental pulp revascularization.
  Interventions: Procedure: intracanal disinfection in revascularization
- Di-antibiotic paste in revascularization (Active Comparator): Revascularization of necrotic anterior teeth: canals disinfection step. Mix 1:1 ciprofloxacin: metronidazole to a final concentration of 0.1 mg/ml, placed as intra-canal medication in the 1st visit of dental pulp revascularization.
  Interventions: Procedure: intracanal disinfection in revascularization

INTERVENTIONS:
Procedure: intracanal disinfection in revascularization — a procedure to create vital cells in the pulp space of immature teeth which enables thickening of the dentinal walls of the root.

SUMMARY:
The object of this study is to compare the effect of Calcium Hydroxide and Di-antibiotic paste as intracanal disinfectants in the 1st visit of revascularization of necrotic immature permanent anterior teeth.

DETAILED DESCRIPTION:
Dental trauma is common in children and it is the main cause of loss of pulp vitality in immature permanent anterior teeth with prevalence rate of 11% and about of 27% of traumatized anterior teeth are left untreated.

Dentists face many challenges during the treatment of infected immature permanent teeth. This is mainly due to the thin dentinal walls of the root and blunderbuss apices that make these teeth susceptible to fracture during and after treatment.

Traditionally, Calcium Hydroxide apexification has been the only method for managing these cases.. however, it was found that this technique caused additional reduction in root strength due to the long-term application of Calcium Hydroxide which may end in fracture of the tooth. The time needed for complete apexification using Calcium Hydroxide was reported to be variable ranging from 5 to 20 months, with failure rate 0f 30% . Therefore, this technique is no longer recommended for the treatment of such cases.

A recently proposed technique for the treatment of immature necrotic permanent teeth is revascularization regenerative endodontic therapy (RET). It is a biologically based technique that allow the continuation of root development and thickening of dentinal walls. This is achieved through proper disinfection o the root canal system, creation of scaffold and perfect coronal seal.

For proper disinfection of the root canal system, antibiotic paste was applied as intracanal dressing for 2-3 weeks. However, the recent recommendations by the European society of Endodontology advices the use of Calcium Hydroxide as intracanal medication instead of intracanal antibiotics. This is because of some concerns regarding the use of antibiotics which include: cytotoxicity to stem cells needed for the revascularization process, risk of antibiotic resistance and the risk of sensitization. Calcium Hydroxide on the other hand is widely used as intracanal disinfectant and some studies were found supporting its use in the revascularization technique, [9, 10]. However, the data available is not sufficient regarding the effectiveness of Calcium Hydroxide in revascularization of necrotic pulp.

Besides, more trials are needed to evaluate the clinical effectiveness of RET in management of immature necrotic permanent teeth as the evidence of using this technique is still weak.

ELIGIBILITY:
Inclusion Criteria:

* Immature anterior teeth with open apices.
* Necrotic teeth (regardless the cause of pulpal involvement: Caries, trauma or congenital anomalies).
* Children free from any systemic diseases that may interfere with the normal healing process.

Exclusion Criteria:

* Children Allergic to antibiotics to be used in the study.
* unooperative children.
* Laxative injuries.
* Compromised remaining tooth structure.
* internal or external root resorption

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Pain | baseline.
  Binary outcome (present/ absent). Assessed by asking the patient
Change in pain | at 6 and 12 months
  Binary outcome (present/ absent). Assessed by asking the patient.

SECONDARY OUTCOMES:
Pain on percussion | baseline and for 1 year follow up
  Binary outcome (present/absent).Assessed by using back of the dental mirror.
Swelling | baseline and for 1 year follow up
  Binary outcome (present/absent). Assessed by visual inspection of labial vestibules.
Sinus or fistula | baseline and for 1 year follow up
  Binary outcome (present/absent). Assessed by visual inspection of labial vestibules.
Root Lengthening | baseline and for 1 year follow up
  Will be evaluated radiographically using DIGORA software. Unit of measurement will be mm.